CLINICAL TRIAL: NCT04367818
Title: Could Peri-anal Block be Effective as Caudal Block in Trans-anal Pull-through Surgery for Children With Hirschsprung Disease??. A Randomized Controlled Trial.
Brief Title: Could Peri-anal Block be Effective as Caudal Block in Trans-anal Pull-through Surgery ??.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Salah Rashed Abd Elraheem, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CPABBEACB
Record Dates: First submitted 2020-04-27; First posted 2020-04-29 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peri-anal local anaesthetic infiltration (Active Comparator): Patients in this group will receive the prepared anesthetic mixture (bupivacaine 0.25% in dose of 1ml\kg plus dexametomidine 2ug\kg diluted in 0.5ml of normal saline) in a syringe will be connected to 22_ gauge short, beveled needle. The technique of the block will be done guided by Nystrom et al.
  Interventions: Procedure: Peri-anal local anaesthetic infiltration
- caudal anaesthesia (Active Comparator): Patients in this group will receive caudal block using 22_gauge short, beveled cannula or needle, The prepared anesthetic mixture (bupivacaine 0.25% in dose of 1ml\kg plus dexametomidine 2ug\kg diluted in 0.5ml of normal saline).
  Interventions: Procedure: Caudal anaesthesia

INTERVENTIONS:
Procedure: Peri-anal local anaesthetic infiltration — postoperative pain relieve, among pediatrics patient
  Arms: Peri-anal local anaesthetic infiltration
Procedure: Caudal anaesthesia — Regional anaesthesia for postoperative pain relieve, among pediatrics patient
  Arms: caudal anaesthesia

SUMMARY:
IN pediatric patient population pain is considered one of the most misunderstood; under diagnosed and under treated medical problems. If left uncontrolled, pain may have a diverse effect on all aspects of life as it is only a sensory perception but also has emotional, cognitive and behavioral components.

DETAILED DESCRIPTION:
Caudal anesthesia is one of the most commonly used regional anesthetic and analgesic technique in pediatric patient as it is an easy safe and reliable method that can be performed for both intraoperative and postoperative analgesia in patient undergoing lower abdominal and lower limb surgery. It can be used for upper abdominal surgery by increasing the volume of local anesthetic injected or through advancing a catheter.

Caudal anesthesia is a common practice given along with general anesthesia to decrease intraoperative inhalational anesthesia requirements, postoperative pain and emergence agitation.

So many patients are complaining from ano-rectal pathologies, these diseases are common in both sexes and all age groups. The spectrum of anorectal disorders ranges from benign and irritating (pruritus- ani) to potentially life-threatening (anorectal cancer) and the surgical intervention is performed mostly under general or regional anesthesia.

While general and regional anesthetics provide reliable anesthesia, they are often associated with nausea,vomiting, urinary retention and motor blockade of lower limbs. Moreover, repeated spinal or epidural punctures performed by inexperienced anesthesiologists often cause delays in the tight schedule of operations.

Several reports have described various forms of local anesthetic infiltration for ano- rectal surgery , hemorrhoidectomy,anal fistula or fissure surgeries or lateral sphincterotomy. Local peri-anal infiltration is a simple procedure that can be easily learned and performed by surgeon and this method allows the operation to begin almost immediately.

There are different types of local anesthesia like infiltration, nerve block, ring block field block. Considering anorectal surgeries, nerve bock mainly pudendal nerve along with infiltration anesthesia is used worldwide. Perianal block by local anesthetic infiltration is safe simple and effective for various anal operations with very high degree of acceptance and satisfaction among patients .it had been found to be associated with low pain score and postoperative complications and faster return to daily social activity.

Although there are studies on the use of caudal block and local infiltration of anesthetic agent for the surgical resolution of anorectal pathologies, there is no established protocol for comparing efficacy, postoperative pain, and satisfaction among pediatrics patient undergoing trans-anal pull through in congenital megacolon (Hirschsprung's disease).

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes.
* Patients with age range 3 to 10 years old.
* Patients with ASA 1 , 2 classification.

Exclusion Criteria:

* Patient or parents refusal.
* Allergy to the study drugs.
* Suspect coagulopathy.
* Local infection at site of intervention.
* History of developmental delay.
* Neuromuscular disorders.
* Skeletal deformity.

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2021-06-30 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Post-operative pain relieve | 24 hours
  Assessment of postoperative pain using FLACC scale and the time to first analgesia request.

SECONDARY OUTCOMES:
Ramsay's sedation scale | 24 hours
  Assessment of postoperative sedation using (Ramsay's sedation scale).
Postoperative motor power | 24 hours
  Assessment of postoperative motor power.
Postoperative Complication | 24 hours
  Assessment of postoperative Complication (nausea, vomiting, bradycardia with heart rate< 80 or hypotension as systolic blood pressure< {70+age in year *2}).

CONTACTS AND LOCATIONS:
Locations (1):
- Mohamed Salah Rashed, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] de Beer DA, Thomas ML. Caudal additives in children--solutions or problems? Br J Anaesth. 2003 Apr;90(4):487-98. doi: 10.1093/bja/aeg064. No abstract available. PMID 12644422
- [Background] Gopal DV. Diseases of the rectum and anus: a clinical approach to common disorders. Clin Cornerstone. 2002;4(4):34-48. doi: 10.1016/s1098-3597(02)90004-9. PMID 12739325
- [Background] Gabrielli F, Cioffi U, Chiarelli M, Guttadauro A, De Simone M. Hemorrhoidectomy with posterior perineal block: experience with 400 cases. Dis Colon Rectum. 2000 Jun;43(6):809-12. doi: 10.1007/BF02238019. PMID 10859082
- [Background] Luck AJ, Hewett PJ. Ischiorectal fossa block decreases posthemorrhoidectomy pain: randomized, prospective, double-blind clinical trial. Dis Colon Rectum. 2000 Feb;43(2):142-5. doi: 10.1007/BF02236970. PMID 10696885
- [Background] Nystrom PO, Derwinger K, Gerjy R. Local perianal block for anal surgery. Tech Coloproctol. 2004 Mar;8(1):23-6. doi: 10.1007/s10151-004-0046-8. PMID 15057585
- [Background] Kaban OG, Yazicioglu D, Akkaya T, Sayin MM, Seker D, Gumus H. Spinal anaesthesia with hyperbaric prilocaine in day-case perianal surgery: randomised controlled trial. ScientificWorldJournal. 2014;2014:608372. doi: 10.1155/2014/608372. Epub 2014 Oct 14. PMID 25379541
- [Background] Zhang Y, Bao Y, Li L, Shi D. The effect of different doses of chloroprocaine on saddle anesthesia in perianal surgery. Acta Cir Bras. 2014 Jan;29(1):66-70. doi: 10.1590/S0102-86502014000100010. PMID 24474180
- [Background] Anannamcharoen S, Cheeranont P, Boonya-usadon C. Local perianal nerve block versus spinal block for closed hemorrhoidectomy: a ramdomized controlled trial. J Med Assoc Thai. 2008 Dec;91(12):1862-6. PMID 19133521